CLINICAL TRIAL: NCT00100386
Title: Strategies to Reduce Transmission of Antimicrobial Resistant Bacteria in Intensive Care Units (STAR*ICU) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 02-081; BAMSG 4-01; NCT00342745 (obsolete NCT alias)
Record Dates: First submitted 2004-12-30; First posted 2004-12-31 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2007-10

CONDITIONS: Bacterial Diseases
Keywords: Hand hygiene, antibiotic resistance, contact precautions
MeSH Terms: conditions — Bacterial Infections

INTERVENTIONS:
Procedure: Intensive Control Strategy
Behavioral: Standard Control Strategy

SUMMARY:
Primary Outcome Measures:Incidence density of colonization with MRSA or VRE (number of new colonization events per 1000 patient days at risk) during the intervention phase. Secondary Outcome Measures:The effect of the 2 strategies on the incidence density of colonization with MRSA and VRE individually will be determined and compared descriptively. The effect of the strategies on the cumulative incidence of bacteremia caused by MRSA and VRE will be determined to assess the clinical relevance of the strategy in preventing infection. The trial will evaluate the frequency of hand hygiene and the use of gloves and gowns by healthcare workers to substantiate whether the effect of the intensive control strategy is mediated, as expected, by an increase in the use of gloves and gowns due to an increase in the number of patients cared for using Contact Precautions.

DETAILED DESCRIPTION:
This study will determine if rates of colonization and infection with 2 resistant Gram positive bacteria-methicillin resistant Staphylococcus aureus (MRSA) and vancomycin resistant enterococci (VRE) among patients in adult intensive care units (ICUs) are lower in ICUs that use an intensive infection control strategy plus standard care compared to ICUs that use standard care alone. The intensive control strategy involves: 1) identifying patients who are colonized with MRSA or VRE by reporting the results of surveillance cultures of the anterior nares and stool or perianal area; 2) Universal Gloving (use of gloves during interactions with the patient or the patient's environment) until the patients are discharged or their surveillance culture results show they are not colonized with MRSA or VRE (whichever happens first); and 3) Contact Precautions (use of gloves and gowns during interactions with the patient or the patient's environment) during care of patients who are colonized with MRSA or VRE. Standard care involves proper hand hygiene (handwashing or use of a waterless hand antiseptic) and use of Standard Precautions (use of gloves and other barriers as needed for interactions involving contact with mucous membranes, wounds, and body fluids) and collection of surveillance cultures, but not reporting of results to these sites. The surveillance cultures will be performed by obtaining swabs of the nose and stool or perianal area from patients upon admission to the ICU, at weekly intervals thereafter, and upon discharge from the ICU. The results of the surveillance cultures will be used to compare the rate of colonization with MRSA and VRE in ICUs using the intensive control strategy with those that use standard care alone.

ELIGIBILITY:
Inclusion Criteria:

ICUs that meet all of the following criteria are eligible to participate in the study:

1. Adult medical, surgical, or medical/surgical ICU, meeting the following descriptions:

   Medical ICU->=80% of patients have medical conditions and have not undergone a surgical procedure during their hospital stay (patients weaned from mechanical ventilation may be included); Surgical ICU->=80% of patients have undergone a surgical procedure during their hospital stay (thoracic, cardiovascular, abdominal, orthopedic, neurosurgical, transplant, urologic, and trauma surgery procedures may be included); and Medical/surgical ICU-a roughly equivalent mixture of patients with medical conditions who have not undergone surgical procedures and patients who have undergone surgical procedures during their hospitalization (i.e., each group constitutes more than 20% and less than 80% of the total number of patients).
2. Patient volume of >=1200 patient days/6 months or >=2400 patient days/12 months during 2002, 2003, or 2004;
3. Incidence density of colonization of >=9 colonization events with either MRSA or VRE/1000 ICU patient days based on results of clinical cultures during 2002, 2003, or 2004;
4. Ability to collect the data required for the analysis;
5. Written approval of the study from the institution's IRB; and
6. Signed protocol signature page indicating willingness to enroll ICU in the study from the ICU physician and the ICU nursing directors.

Exclusion Criteria:

Intensive care units that meet any of the following criteria are excluded from the study:

1. Coronary care, burn, bone marrow/hematopoetic stem cell transplant, neurosurgical, pediatric, or neonatal ICUs;
2. ICUs currently screening all patients for colonization with MRSA and VRE on admission to the ICU and at least once a week during their ICU stay with results of surveillance cultures reported to clinicians (Note: ICUs screening only selected, "high-risk" patients, screening patients on admission to the ICU but not an ongoing basis, or screening patients for MRSA or VRE but not both MRSA and VRE are not excluded);
3. ICUs currently with a policy for Universal Gloving for all patient contact regardless of whether the patient is known to be colonized with VRE or MRSA;
4. ICUs planning to enroll subjects in studies testing investigational agents administered for the purpose of eradicating or preventing colonization with MRSA or VRE or devices or practice management strategies that have colonization and/or infection with resistant organisms as an outcome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30000
Dates: Start 2005-03; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Yale University, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Cooper University Hospital, Camden, New Jersey
  - Beth Israel Medical Center, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon

REFERENCES:
- [Result] Huskins WC, Huckabee CM, O'Grady NP, Murray P, Kopetskie H, Zimmer L, Walker ME, Sinkowitz-Cochran RL, Jernigan JA, Samore M, Wallace D, Goldmann DA; STAR*ICU Trial Investigators. Intervention to reduce transmission of resistant bacteria in intensive care. N Engl J Med. 2011 Apr 14;364(15):1407-18. doi: 10.1056/NEJMoa1000373. PMID 21488763